CLINICAL TRIAL: NCT03042546
Title: Calcium Sulfate Spacer in Open Tibia Fractures With Sub-segmental Bone Loss to Decrease the Need for Secondary Surgery
Brief Title: Calcium Sulfate Spacer in Open Tibia Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention. Low enrollment and PI leaving institution
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Claude Sagi, Professor, Orthopedics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002348
Record Dates: First submitted 2017-01-27; First posted 2017-02-03 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Open tíbia Fracture With Sub-segmental Bone Loss
MeSH Terms: interventions — Calcium Sulfate; Polymethyl Methacrylate

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calcium Sulphate (Active Comparator)
  Interventions: Drug: Calcium Sulfate
- PMMA (Active Comparator)
  Interventions: Drug: PMMA
- Nothing (Active Comparator)
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Calcium Sulfate — Calcium Sulfate with abx will be used in the defect
  Arms: Calcium Sulphate
Drug: PMMA — PMMA with abx will be used in the defect
  Arms: PMMA
Other: No treatment — The defect will not be treated
  Arms: Nothing

SUMMARY:
Investigators will compare antibiotic impregnated Calcium sulfate versus PMMA versus nothing in these sub-segmental bone defects.

ELIGIBILITY:
Inclusion Criteria:

* Open tibia shaft fracture treated with an IMN

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Sagi, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
there is no plan to share individual data

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only enrolled patient was not randomized
Period: Overall Study
Arm/Group | Calcium Sulphate | PMMA | Nothing
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: project abandoned
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcium Sulphate | PMMA | Nothing | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Nonunion
Description: Radiographic healing at one year with no additional surgery
Time Frame: One Year
Population: project was abandoned as PI left institution
Arm/Group | Calcium Sulphate | PMMA | Nothing
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: no one randomized or treated
Arm/Group | Calcium Sulphate | PMMA | Nothing
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT03042546/Prot_SAP_000.pdf